CLINICAL TRIAL: NCT02557815
Title: Changing the Vulnerable Brain: A Neuromodulation Study in Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Anneke E. Goudriaan, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EA1027; 91713354 (Other Grant/Funding Number: Dutch Scientific Foundation (ZonMw)); EA1027 (Other Grant/Funding Number: The European Foundation for Alcohol Research (ERAB))
Record Dates: First submitted 2015-09-06; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Alcohol Dependence
Keywords: Repetitive Transcranial Magnetic Stimulation; Emotion Regulation; Craving
MeSH Terms: conditions — Alcoholism; Emotional Regulation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): Repetitive Transcranial Magnetic Stimulation: Active 10hz stimulation over the right dorsolateral Prefrontal Cortex (dlPFC)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham stimulation (Sham Comparator): Repetitive Transcranial Magnetic Stimulation: sham stimulation over the right dlPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive 10Hz right DLPFC stimulation using Magstim TMS apparatus

SUMMARY:
This current project investigates the effect of a single session of right dlPFC repetitive transcranial magnetic stimulation on emotion regulation abilities and craving in alcohol dependent patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependence
* Currently abstinent

Exclusion Criteria:

* psychoactive medication
* not eligible for MRI (metals or claustrophobia)
* (familial) history of epilepsy
* current psychiatric disorders (besides alcohol dependence)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in BOLD response during an emotion regulation task (fMRI) | Change in BOLD response from baseline, compared to BOLD response after stimulation (approximately two weeks later)
  BOLD response was measured during an emotion regulation task. The change in BOLD response between sessions is the primary outcome for this study

SECONDARY OUTCOMES:
Change in experienced emotion during an emotion regulation task with Visual Analogue Scales (VAS) | Change in experienced emotion from baseline, and after the stimulation session (approximately two weeks later)
  Participants were instructed to either 'attend' or 'regulate' their emotion associated with the presented (negatively valenced) pictures. Experienced (or regulated) emotion was assessed with visual analogue scales (VAS).
Change in craving levels [Alcohol Urge Questionnaire (AUQ)] | Before and after the emotion regulation task, during both baseline and stimulation session (e.g. 4 time points, sessions were separated by approximately two weeks)
  The AUQ was administered in order to assess craving levels. The AUQ consists of eight statements wich are rated on a 7 point likert scale [0 = Strongly disagree, 6 = Strongly Agree]

CONTACTS AND LOCATIONS:
Overall Officials: Anneke E Goudriaan, Prof dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

REFERENCES:
- [Background] Jansen JM, van Holst RJ, van den Brink W, Veltman DJ, Caan MW, Goudriaan AE. Brain function during cognitive flexibility and white matter integrity in alcohol-dependent patients, problematic drinkers and healthy controls. Addict Biol. 2015 Sep;20(5):979-89. doi: 10.1111/adb.12199. Epub 2014 Dec 5. PMID 25477246
- [Result] Jansen JM, Daams JG, Koeter MW, Veltman DJ, van den Brink W, Goudriaan AE. Effects of non-invasive neurostimulation on craving: a meta-analysis. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2472-80. doi: 10.1016/j.neubiorev.2013.07.009. Epub 2013 Jul 31. PMID 23916527
- [Derived] Jansen JM, van den Heuvel OA, van der Werf YD, de Wit SJ, Veltman DJ, van den Brink W, Goudriaan AE. The Effect of High-Frequency Repetitive Transcranial Magnetic Stimulation on Emotion Processing, Reappraisal, and Craving in Alcohol Use Disorder Patients and Healthy Controls: A Functional Magnetic Resonance Imaging Study. Front Psychiatry. 2019 May 7;10:272. doi: 10.3389/fpsyt.2019.00272. eCollection 2019. PMID 31133889
- [Derived] Jansen JM, van den Heuvel OA, van der Werf YD, de Wit SJ, Veltman DJ, van den Brink W, Goudriaan AE. Emotion Processing, Reappraisal, and Craving in Alcohol Dependence: A Functional Magnetic Resonance Imaging Study. Front Psychiatry. 2019 Apr 9;10:227. doi: 10.3389/fpsyt.2019.00227. eCollection 2019. PMID 31057439